CLINICAL TRIAL: NCT01580397
Title: A Multicenter, Phase 2 Study to Investigate the Preliminary Efficacy and Safety of INNO-206 in Subjects With Advanced or Unresectable Pancreatic Ductal Carcinoma Whose Tumors Have Progressed Following Prior Treatment
Brief Title: Pilot Phase 2 Study to Investigate the Preliminary Efficacy and Safety of INNO-206 in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-206-P2-PDA-01
Record Dates: First submitted 2012-04-13; First posted 2012-04-19 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2013-06

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic cancer; INNO-206; Doxorubicin-EMCH
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — DOXO-EMCH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- INNO-206 (Experimental): INNO-206 administered at 350 mg/m2 (260 mg/m2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 8 consecutive cycles.
  Interventions: Drug: INNO-206

INTERVENTIONS:
Drug: INNO-206 — INNO-206 at a total dose of 350 mg/m2 (260 mg/m2 doxorubicin equivalent) will be administered as a 30 minute IV infusion every 21 days.
  Other Names: Aldoxorubicin

SUMMARY:
Patients with metastatic, locally advanced, or unresectable pancreatic ductal carcinomas (PDA) who have failed prior chemotherapy with gemcitabine regimens have an extremely poor prognosis with progression-free survival of around 13 weeks and median overall survival of approximately 20 weeks after second line chemotherapy. Recent studies suggest that albumin may be preferentially concentrated in pancreatic cancers that appear to be starved for this protein. Thus, any molecule attached to albumin would also collect inside the tumor. Based on its postulated mechanism of action, INNO-206 may improve the activity of doxorubicin without increasing its toxicity, as has been demonstrated in animal studies, and induce enhanced anti-tumor efficacy.

DETAILED DESCRIPTION:
This is a phase 2 open-label, pilot study evaluating the preliminary efficacy and safety of INNO-206 administered at 350 mg/m2 (260 mg/m2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 8 consecutive cycles.

Tumor response (complete and partial response and stable disease) will be monitored at Screening, then prior to cycles 3, 5 and 7, 3 weeks after cycle 8, then every 2 months to month 8 and every 3 months to tumor progression using the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria, and treatment will continue every 21 days until tumor progression is observed, 8 cycles of treatment are completed or unacceptable toxicity occurs. Progression-free survival [PFS], stable disease at 4 months and overall survival [OS] will be monitored as other primary objectives. PET/CT will be performed at Baseline and Week 9 to determine change in tumor metabolic activity, and CA 19-9 will be determined serially to assess potential tumor reduction. Subjects will visit the study site every 21 days for their IV infusions, at which time safety monitoring, including AEs, a directed physical examination, laboratory evaluations (serum chemistry, complete blood count [CBC], and urinalysis), vital signs, weight measurements, ECOG performance status and ECGs will be performed. Cardiac function will also be followed periodically using ECHOs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age; male or female.
* Histologically or cytologically confirmed, locally advanced, unresectable, and/or metastatic pancreatic ductal adenocarcinoma.
* Cancer progression after treatment with one gemcitabine and one fluoropyrimidine-containing chemotherapy regimen.
* Capable of providing informed consent and complying with trial procedures.
* ECOG performance status 0-1.
* Life expectancy ≥ 8 weeks.
* Measurable tumor lesions according to RECIST 1.1 criteria.
* Women must not be able to become pregnant (eg post-menopausal for at least 1 year, surgically sterile, or practicing adequate birth control methods) for the duration of the study. (Adequate contraception includes: oral contraception, implanted contraception, intrauterine device implanted for at least 3 months, or barrier method in conjunction with spermicide.)
* Women of child bearing potential must have a negative serum or urine pregnancy test at the Screening Visit and be non-lactating.
* Geographic accessibility to the site.

Exclusion Criteria:

* Prior exposure to > 3 cycles or 225 mg/m2 of doxorubicin or Doxil®.
* Palliative surgery and/or radiation treatment less than 4 weeks prior to Randomization.
* Exposure to any investigational agent within 30 days of Randomization.
* Evidence of central nervous system (CNS) metastasis (negative imaging study, if clinically indicated, within 4 weeks of Screening Visit).
* History of other malignancies (except cured basal cell carcinoma, superficial bladder cancer or carcinoma in situ of the cervix) unless documented free of cancer for ≥ 5 years.
* Laboratory values: Screening serum creatinine > 1.5x upper limit of normal (ULN), alanine aminotransferase (ALT) > 3×ULN or > 5×ULN if liver metastases are present, total bilirubin > 3×ULN, absolute neutrophil count < 1,500/mm3, platelet concentration < 100,000/mm3, absolute lymphocyte count < 1000/mm3, hematocrit level < 27% for females or < 30% for males, or coagulation tests (prothrombin time [PT], partial thromboplastin time [PTT], International Normalized Ratio [INR]) > 1.5×ULN, serum albumin ≤ 2.8 g/dL.
* Clinically evident congestive heart failure > class II of the New York Heart Association (NYHA) guidelines.
* Current, serious, clinically significant cardiac arrhythmias, defined as the existence of an absolute arrhythmia or ventricular arrhythmias classified as Lown III, IV or V.
* History or signs of active coronary artery disease with or without angina pectoris.
* Serious myocardial dysfunction ultrasound-determined, with absolute left ventricular ejection fraction (LVEF) < 45% of predicted.
* History of HIV infection.
* Active, clinically significant serious infection requiring treatment with antibiotics, anti-virals or anti-fungals.
* Major surgery within 4 weeks prior to Randomization.
* Substance abuse or any condition that might interfere with the subject's participation in the study or in the evaluation of the study results.
* Any condition that is unstable and could jeopardize the subject's participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-05-16 (Actual); Primary Completion 2013-05-13 (Actual); Study Completion 2013-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Von Hoff, MD, FACP, Principal Investigator — Translational Genomics Research Institute; Daniel Levitt, MD, PhD, Study Director — CytRx
Locations (6):
- United States (6):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - Sarcoma Oncology Center, Santa Monica, California
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Medical College of Wisconsin - Division of Neoplastic Diseases and Related Disorders, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 subjects were enrolled, whereas 14 subjects participated.
  1 subject died prior to treatment start and was not included in analysis.
Period: Overall Study
Arm/Group | INNO-206
Started | 14
Completed | 0
Not Completed | 14
Not completed — Lack of Efficacy | 14

BASELINE CHARACTERISTICS:
Population: Those subjects that received at least one dose of INNO-206.
Groups:
- INNO-206: INNO-206 administered at 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 8 consecutive cycles.
Arm/Group | INNO-206
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (4.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Subjects with Advanced or Unresectable Pancreatic Ductal Carcinoma [Count of Participants; unit: Participants] | 15

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective responses were evaluated using the Response Evaluation Criteria In Solid Tumors 1.1 (RECIST 1.1). Changes (ie, improvements) in tumor measurements from baseline values were assigned a status of CR or PR or SD. Objective response measurements comprised the sum of CR plus PR.
  Complete Response (CR): disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm).
  Partial Response (PR): >=30% decrease in the sum of the longest diameter of target lesions, from the baseline sum longest diameter.
Time Frame: Approximately 12 months from enrollment
Population: These subjects had more than one cycle of treatment and/or were able to be evaluated for response or disease progression.
Measure: Count of Participants; unit: Participants
Groups:
- INNO-206: INNO-206 administered at 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) intravenously (IV) on Day 1 every 21 days for up to 8 consecutive cycles.
  INNO-206: INNO-206 at a total dose of 350 mg/m^2 (260 mg/m^2 doxorubicin equivalent) will be administered as a 30 minute IV infusion every 21 days.
Arm/Group | INNO-206
Number analyzed (Participants) | 9
Participants | 0

2. Secondary Outcome: Number of Participants With Treatment-related Toxicities (Adverse Events)
Description: The primary objective of this study is to determine the preliminary safety of administration of aldoxorubicin in subjects with advanced or unresectable pancreatic ductal adenocarcinoma as measured by the frequency and severity of adverse events (AEs).
  The following assessments were used to determine if subjects had adverse events:
  vitals signs (systolic/diastolic blood pressure, pulse, respiration, temperature, weight, and body surface area) physical examination laboratory tests (chemistry, hematology, urinalysis, BSA) additionally, the following scans were performed to determine adverse events: ECHO / MUGA ECG
Time Frame: 30 days after last dose, up to 178 days
Measure: Count of Participants; unit: Participants
Arm/Group | INNO-206
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) that occurred after any administration of the study medication were to be followed until the event resolved, until the subject began alternative treatment, or until the end of the study. All SAEs that occurred during the course of the study or within 30 days of the last administration of study medication were to be reported, up to 178 days.
Description: 1 participant signed consent, but did not receive first dose. That subject died.
Arm/Group | INNO-206
All-Cause Mortality (participants affected / at risk) | 13/15
Serious Adverse Events (participants affected / at risk) | 11/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INNO-206 (N=14)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 1
Rectal obstruction (Gastrointestinal disorders) | 1
Small intestine obstruction (Gastrointestinal disorders) | 2
Diverticulitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Influenza-Stomach (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic event (Vascular disorders) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INNO-206 (N=14)
Anemia (Blood and lymphatic system disorders) | 4
Febrile Neutropenia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 2
Gastrointestinal disorders, other (Gastrointestinal disorders) | 2
Gastrointestinal pain (Gastrointestinal disorders) | 1
Mucositis oral (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 6
Rectal obstruction (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 11
Fever (General disorders) | 3
Gait disturbance (General disorders) | 1
Infections and infestations, other (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 11
Platelet count decreased (Investigations) | 4
Weight loss (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Ataxia (Nervous system disorders) | 1
Concentration impairment (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1
Stroke (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal and urinary disorder- other (Renal and urinary disorders) | 1
Urinary frequency (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thromboembolic event (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-04-03): https://cdn.clinicaltrials.gov/large-docs/97/NCT01580397/Prot_SAP_000.pdf